CLINICAL TRIAL: NCT03624257
Title: Comparing Two Treatment Modalities of Peri-implantitis - Blue Laser (445 nm) and Conventional Flap Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision: priority change (Study approved by ethics committee and Swedish competent authority)
Sponsor: Sirona Dental Systems GmbH (Industry)
Responsible Party: Principal Investigator, Annsofi Johannsen, Registered Dental Hygienist (RDH); Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Peri-implantitis 445 nm laser; CIV-1 8-06-024304 (Other: EUDAMED)
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Peri-Implantitis
Keywords: Laser treatment; surgical treatment; patient reported outcomes; microbiology; immunology; radiological examination
MeSH Terms: conditions — Peri-Implantitis | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Masking for the assessors of microbial, immunological and radiographic analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scaling and root planning + Laser treatment (Experimental)
  Interventions: Device: Laser treatment
- Mucosal flap surgery (Active Comparator)
  Interventions: Procedure: Mucosal flap surgery

INTERVENTIONS:
Device: Laser treatment — The participants in the laser group are treated by a combination of scaling and root planning (SRP) and 445 nm diode laser. The peri-implant pocket will be radiated with the 445 nm laser, removing bacteria, diseased epithelium and granulation tissue. The Power setting on the laser will be 0.7 W continuous wave and will be used at maximum 20 s Before cooling water is applied. Total treatment time will vary with the depth of the pocket and size of the surrounding bone crater.
  Arms: Scaling and root planning + Laser treatment
Procedure: Mucosal flap surgery — The participants will receive a conventional peri-implant mucosal flap surgery of affected implants, in combination with scaling and root planning (SRP), and return after 7-10 days for suture removal. The surgery is a well-established treatment of peri-implantitis.
  Arms: Mucosal flap surgery

SUMMARY:
A clinical trial comparing laser treatment and conventional mucosal flap surgery for treatment of peri-implantitis. The main aim of the study is to evaluate if treatment of peri-implantitis with a novel blue laser (445 nm) combined with scaling and root planning (SRP) is clinically comparable to conventional mucosal flap surgery in terms of pocket probing depth reduction.

DETAILED DESCRIPTION:
The present project aims to evaluate a novel method in treating peri-implantitis, with focus on decreasing the patient's suffering as well as disease progression. Peri-implantitis has a direct influence on both physical and psychological well-being and have been related to difficulty in chewing due to loss of implants, bad esthetic appearance as well as high costs. Therefore, it is of importance for the individual as well as for the society to thoroughly investigate any new treatment approaches.

The study is a prospective randomized clinical trial comparing laser treatment (test group) and conventional mucosal flap surgery (active control group). Assessment of clinical variables at baseline and after 6 months. Patient reported outcomes at baseline, directly after treatment and after 10 days.

Primary Objective:

To evaluate if treatment of peri-implantitis with a novel blue laser (445 nm) combined with scaling and root planning (SRP) is clinically comparable to conventional mucosal flap surgery in terms of pocket probing depth reduction.

Secondary Objectives:

* To evaluate other clinical and radiological variables connected to peri-implantitis and the inflammation surrounding the dental implant.
* To evaluate the patient experience of a novel blue laser for treatment of peri-implantitis.
* To evaluate the inflammatory and microbial response after laser treatment

ELIGIBILITY:
Inclusion Criteria:

* Signs of peri-implantitis around one or more dental implants. All criteria below need to be fulfilled for inclusion.

  * Presence of pocket probing depth (PPD) > 5 mm
  * Bleeding on probing/suppuration (BOP/Pus)
  * At least 2 mm loss of bone, visible on radiographs, after initial osseointegration.
* ≥ 18 years old.
* Patient able to understand Swedish.

Exclusion Criteria:

* Antibiotic treatment 6 months prior to baseline.
* Peri-implant treatment 6 months prior to baseline.
* Myocardial infarction 6 months prior to baseline.
* Previous radiation treatment in the affected jaw area.
* Previous i.v. bisphosphonate treatment.
* Moderate or severe impairment of cognitive function (e.g. dementia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in Pocket probing depth (PPD) at 6 months after treatment. | At baseline and 6 months post treatment
  Pocket probing depth (PPD) will be measured by a 1 mm graded pocket probe from the bottom of the peri-implant pocket to the marginal mucosa and will be registered on 4 surfaces surrounding the implant.

SECONDARY OUTCOMES:
Mean change from baseline in Plaque index (PI) at 6 months after treatment. | At baseline and 6 months post treatment
  Plaque index (PI) will be measured at 4 sites per implant and assessed as per cent of the total amount of measured implant surfaces.
Mean change from baseline in Bleeding on probing (BOP) at 6 months after treatment. | At baseline and 6 months post treatment
  BOP will be registered on 4 surfaces surrounding the implant after probing the peri-implant pocket with a pocket probe, up to 20 s after the provocation with the probe.
Mean change from baseline in Recession of the marginal mucosa at 6 months after treatment. | At baseline and 6 months post treatment
  Recession of the marginal mucosa will be measured from a per implant decided fixed point like the shoulder of the implant or the edge of the prosthetic to the marginal mucosa. Registered on 4 surfaces surrounding the implant.
Mean change from baseline in Presence of suppuration at 6 months after treatment. | At baseline and 6 months post treatment
  Presence of suppuration will be registered on 4 surfaces surrounding the implant after probing the peri-implant pocket with a pocket probe, up to 20 s after the provocation with the probe.
Mean change from baseline in Marginal bone level on radiographs at 6 months after treatment. | At baseline and 6 months post treatment
Mean change from baseline in Patient reported outcome using the VAS score directly post treatment. | At baseline and immediately post treatment.
  Visual analogue scale (VAS) is used to record the patients pain, discomfort and satisfaction with the treatment.
Mean change from baseline in Patient reported outcome using the VAS score at 10 days post treatment. | At baseline and 10 days post treatment.
  Visual analogue scale (VAS) is used to record the patients pain, discomfort and satisfaction with the treatment.
Mean change from baseline in the inflammatory response in the inflammatory exudates at 6 months after treatment. | At baseline and 6 months post treatment
  Analysis of inflammatory meditators in gingival crevicular fluid (GCF) and saliva will be performed by commercially available ELISAs or multiplex assays.
Bacterial composition of the subgingival microflora | At baseline and 6 months post treatment
  The bacterial composition in the subgingival microflora will be analyzed by quantitative real-time Polymerase Chain Reaction (qPCR).

CONTACTS AND LOCATIONS:
Overall Officials: Annsofi Johannsen, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Danakliniken Specialist Dentistry, Mörby Centrum floor 5, Danderyd
  - Specialist Dentistry Clinic, Karolinska Institutet, Dept. of Dental Medicine, Karolinska Institutet, Huddinge

IPD SHARING:
Plan to Share IPD: No